CLINICAL TRIAL: NCT00639938
Title: A Phase III Randomized Clinical Trial of the Standard Two Dose Nevirapine (NVP) Regimen With the Addition of HIV Immune Globulin(HIVIGLOB) or Extended Infant NVP Dosing Compared With the Standard NVP Regimen Alone for the Prevention of Maternal-Infant HIV Transmission in Uganda
Brief Title: Nevirapine Study for the Prevention of Maternal-Infant HIV Transmission in Uganda
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Brooks Jackson, MD, Johns Hopkins School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01AI034235 (NIH)
Record Dates: First submitted 2008-03-18; First posted 2008-03-20 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: HIV Infections
Keywords: Pregnancy, High-Risk; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Mother dosing regimen: Single dose of 200 mg NVP taken orally at onset of labor
  Infant dosing regimen: Single dose of 2 mg/kg NVP taken orally within the first week after delivery
  Interventions: Drug: Nevirapine
- 2 (Experimental): Mother dosing regimen: Single dose of 200 mg NVP taken orally at onset of labor
  Infant dosing regimen: 2 mg/kg NVP taken orally within the first week after delivery and 5 mg NVP taken orally daily from Day 8 through Week 6
  Interventions: Drug: Nevirapine
- 3 (Experimental): Mother dosing regimen: Single 12 gm intravenous dose of HIVIGLOB at 36 - 37 weeks gestation and 200 mg NVP taken orally at onset of labor
  Infant dosing regimen: Single 1.2 gm intravenous dose HIVIGLOB within 18 hours of birth and 2 mg/kg NVP taken orally within the first week after delivery
  Interventions: Drug: Nevirapine; Drug: HIV immune globulin solution

INTERVENTIONS:
Drug: Nevirapine — 200 mg Nevirapine tablet
  Other Names: NVP Viramune
Drug: HIV immune globulin solution — 5% intravenous HIV immune globulin solution
  Other Names: HIVIGLOB
  Arms: 3

SUMMARY:
The increase in pediatric HIV infection has a substantial impact on childhood mortality in the developing world. A number of recent studies suggest that as many as half or more of mother-to-child HIV transmissions in developing countries occur in late pregnancy or during labor and delivery. Interventions targeted during the perinatal period have shown to be effective and to have a significant impact in reducing transmission. The purpose of this study is to investigate the effectiveness of nevirapine (NVP) plus immunoprophylaxis or extended NVP dosing regimens in HIV-infected pregnant women and their infants during the perinatal period.

DETAILED DESCRIPTION:
There is an urgent need to find safe, effective means of preventing mother-to-child-transmission (MTCT) of HIV that can be used in developing countries. One of the greatest obstacles to prevention in these areas remains HIV transmission through breast milk. The primary purpose of this trial is to determine if nevirapine (NVP) plus immunoprophylaxis (by intravenous HIV immune globulin [HIVIGLOB]) or extended NVP dosing of the neonate during the perinatal period can safely and effectively reduce the risk of peripartum or early breastfeeding-related HIV MTCT.

This study will last 11-18 weeks for each mother and 18 months for each infant. HIV-infected pregnant women will be randomly assigned to one of three arms. Participants in Arm 1 will receive a single dose of 200 mg NVP orally at the onset of labor. Infants in Arm 1 will receive a single dose of 2 mg/kg NVP orally within the first week after delivery. Arm 2 participants will receive a single dose of 200 mg NVP orally at the onset of labor. Infants in Arm 2 will receive 2 mg/kg NVP orally within the first week after delivery and 5 mg NVP taken orally daily from Day 8 through Week 6. Arm 3 participants will receive a 12 gm intravenous dose of HIVIGLOB at 36-37 weeks gestation and 200 mg NVP orally at the onset of labor. Infants in Arm 3 will receive a single 1.2 gm intravenous dose HIVIGLOB within 18 hours of birth and 2 mg/kg NVP orally within the first week after delivery.

There will be five or six study visits for pregnant participants. A targeted medical history, physical examination, and blood collection will occur at all visits. After birth, there will be 11 study visits for infants in Arms 1 and 2 and 12 study visits for infants in Arm 3. Medical history and a targeted physical exam will occur at all visits. Blood collection will occur at some visits.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant between 32-36 weeks estimated gestation
* HIV Infected
* Intent to breastfeed infant
* Certain laboratory criteria. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Sensitivity to immune globulin preparations or any benzodiazepine
* Clinically significant disease, as determined by the investigator, that would compromise the ability of the participant to complete the study requirements
* Currently receiving antiretroviral therapy (other than the intrapartum NVP or other peripartum regimens)
* Participation in any HIV vaccine trials
* History of cytotoxic chemotherapy within one month of study entry
* Uncontrolled hypertension
* Chronic alcohol or illicit drug use
* History of non-compliance with visits or medication
* Women who become pregnant again during study follow-up will not be eligible for re-enrollment in the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2004-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Rate of HIV infection in infants born to study participants in each arm of the study | At Birth, Weeks 2, 6, and 14, and Months 6, 12, and 18
Safety and tolerance of HIVIGLOB given to pregnant women at 36-37 weeks gestation and neonates at birth in combination with NVP and of NVP alone | Throughout study

SECONDARY OUTCOMES:
Rate of immunologic progression in HIV-infected infants in each arm | Throughout study
Infant mortality | Throughout study
Maternal plasma HIV RNA levels at delivery | At Birth
Immunologic, virologic, and pharmacologic factors | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Brooks Jackson, MD, Principal Investigator — Johns Hopkins School of Medicine

REFERENCES:
- [Background] Colvin M, Chopra M, Doherty T, Jackson D, Levin J, Willumsen J, Goga A, Moodley P; Good Start Study Group. Operational effectiveness of single-dose nevirapine in preventing mother-to-child transmission of HIV. Bull World Health Organ. 2007 Jun;85(6):466-73. doi: 10.2471/blt.06.033639. PMID 17639244
- [Background] Flys TS, Mwatha A, Guay LA, Nakabiito C, Donnell D, Musoke P, Mmiro F, Jackson JB, Eshleman SH. Detection of K103N in Ugandan women after repeated exposure to single dose nevirapine. AIDS. 2007 Oct 1;21(15):2077-82. doi: 10.1097/QAD.0b013e3282703847. PMID 17885298
- [Background] Jackson JB, Musoke P, Fleming T, Guay LA, Bagenda D, Allen M, Nakabiito C, Sherman J, Bakaki P, Owor M, Ducar C, Deseyve M, Mwatha A, Emel L, Duefield C, Mirochnick M, Fowler MG, Mofenson L, Miotti P, Gigliotti M, Bray D, Mmiro F. Intrapartum and neonatal single-dose nevirapine compared with zidovudine for prevention of mother-to-child transmission of HIV-1 in Kampala, Uganda: 18-month follow-up of the HIVNET 012 randomised trial. Lancet. 2003 Sep 13;362(9387):859-68. doi: 10.1016/S0140-6736(03)14341-3. PMID 13678973
- [Derived] Onyango-Makumbi C, Omer SB, Mubiru M, Moulton LH, Nakabiito C, Musoke P, Mmiro F, Zwerski S, Wigzell H, Falksveden L, Wahren B, Antelman G, Fowler MG, Guay L, Jackson JB. Safety and efficacy of HIV hyperimmune globulin for prevention of mother-to-child HIV transmission in HIV-1-infected pregnant women and their infants in Kampala, Uganda (HIVIGLOB/NVP STUDY). J Acquir Immune Defic Syndr. 2011 Dec 1;58(4):399-407. doi: 10.1097/QAI.0b013e31822f8914. PMID 21826009
- [Derived] Six Week Extended-Dose Nevirapine (SWEN) Study Team; Bedri A, Gudetta B, Isehak A, Kumbi S, Lulseged S, Mengistu Y, Bhore AV, Bhosale R, Varadhrajan V, Gupte N, Sastry J, Suryavanshi N, Tripathy S, Mmiro F, Mubiru M, Onyango C, Taylor A, Musoke P, Nakabiito C, Abashawl A, Adamu R, Antelman G, Bollinger RC, Bright P, Chaudhary MA, Coberly J, Guay L, Fowler MG, Gupta A, Hassen E, Jackson JB, Moulton LH, Nayak U, Omer SB, Propper L, Ram M, Rexroad V, Ruff AJ, Shankar A, Zwerski S. Extended-dose nevirapine to 6 weeks of age for infants to prevent HIV transmission via breastfeeding in Ethiopia, India, and Uganda: an analysis of three randomised controlled trials. Lancet. 2008 Jul 26;372(9635):300-13. doi: 10.1016/S0140-6736(08)61114-9. PMID 18657709